CLINICAL TRIAL: NCT04333550
Title: Application of Iron Chelator (Desferal) to Reduce the Severity of COVID-19 Manifestations
Brief Title: Application of Desferal to Treat COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kermanshah University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Yadollah Shakiba, Dr. Yadollah Shakiba, MD, PhD, Kermanshah University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1398.1224
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: COVID-19, Deferoxamine
MeSH Terms: conditions — COVID-19 | interventions — Deferoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Desferal addition to standard treatment (Experimental)
  Interventions: Drug: Deferoxamine
- Experimental: standard treatment (Experimental)
  Interventions: Drug: Deferoxamine

INTERVENTIONS:
Drug: Deferoxamine — Intravenous infusion of Deferoxamine

SUMMARY:
In this study, defined cases of COVID-19 with mild, moderate or severe pneumonia will be treated with standard treatment regimens in combination with IV injection of Deferoxamine. Improvement in clinical, laboratory and radiological manifestations will be evaluated in treated patient compared to control group.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of COVID-19 Disease,

Exclusion Criteria:

Previous history of allergy to Deferoxamin, Pregnancy, kidney dysfunction,

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | up to 20 days
  All cause of death

SECONDARY OUTCOMES:
change in patients clinical manifestation | up to 20 days
  Mild, Moderate or Severe
change in patients PaO2 | up to 20 days
Length of hospitalization | up to 20 days
  days
C-reactive protein | up to 20 days
lymphocyte count | up to 20 days
length of intensive care unit stay | 1 to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Yadollah Shakiba, MD, PhD, Study Director — Regenerative Medicine Research Center, Kermanshah University of Medical Sciences, Kermanshah, Iran; Amir Kiani, PhD, Principal Investigator — Regenerative Medicine Research Center, Kermanshah University of Medical Sciences, Kermanshah, Iran
Locations (1):
- Regenerative Medicine Research Center, Kermanshah University of Medical Sciences, Kermanshah, Iran, Kermanshah, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Drakesmith H, Prentice A. Viral infection and iron metabolism. Nat Rev Microbiol. 2008 Jul;6(7):541-52. doi: 10.1038/nrmicro1930. PMID 18552864
- [Result] Nairz M, Haschka D, Demetz E, Weiss G. Iron at the interface of immunity and infection. Front Pharmacol. 2014 Jul 16;5:152. doi: 10.3389/fphar.2014.00152. eCollection 2014. PMID 25076907
- [Result] Georgiou NA, van der Bruggen T, Oudshoorn M, Nottet HS, Marx JJ, van Asbeck BS. Inhibition of human immunodeficiency virus type 1 replication in human mononuclear blood cells by the iron chelators deferoxamine, deferiprone, and bleomycin. J Infect Dis. 2000 Feb;181(2):484-90. doi: 10.1086/315223. PMID 10669330
- [Result] Vlahakos D, Arkadopoulos N, Kostopanagiotou G, Siasiakou S, Kaklamanis L, Degiannis D, Demonakou M, Smyrniotis V. Deferoxamine attenuates lipid peroxidation, blocks interleukin-6 production, ameliorates sepsis inflammatory response syndrome, and confers renoprotection after acute hepatic ischemia in pigs. Artif Organs. 2012 Apr;36(4):400-8. doi: 10.1111/j.1525-1594.2011.01385.x. Epub 2011 Dec 21. PMID 22187937
- [Result] Wang H, Li Z, Niu J, Xu Y, Ma L, Lu A, Wang X, Qian Z, Huang Z, Jin X, Leng Q, Wang J, Zhong J, Sun B, Meng G. Antiviral effects of ferric ammonium citrate. Cell Discov. 2018 Mar 27;4:14. doi: 10.1038/s41421-018-0013-6. eCollection 2018. PMID 29619244
- [Result] Cinatl J Jr, Cinatl J, Rabenau H, Gumbel HO, Kornhuber B, Doerr HW. In vitro inhibition of human cytomegalovirus replication by desferrioxamine. Antiviral Res. 1994 Sep;25(1):73-7. doi: 10.1016/0166-3542(94)90095-7. PMID 7811060
- [Result] Visseren F, Verkerk MS, van der Bruggen T, Marx JJ, van Asbeck BS, Diepersloot RJ. Iron chelation and hydroxyl radical scavenging reduce the inflammatory response of endothelial cells after infection with Chlamydia pneumoniae or influenza A. Eur J Clin Invest. 2002 Mar;32 Suppl 1:84-90. doi: 10.1046/j.1365-2362.2002.0320s1084.x. PMID 11886437
- [Result] Sappey C, Boelaert JR, Legrand-Poels S, Forceille C, Favier A, Piette J. Iron chelation decreases NF-kappa B and HIV type 1 activation due to oxidative stress. AIDS Res Hum Retroviruses. 1995 Sep;11(9):1049-61. doi: 10.1089/aid.1995.11.1049. PMID 8554902
- [Result] Chang HC, Bayeva M, Taiwo B, Palella FJ Jr, Hope TJ, Ardehali H. Short communication: high cellular iron levels are associated with increased HIV infection and replication. AIDS Res Hum Retroviruses. 2015 Mar;31(3):305-12. doi: 10.1089/aid.2014.0169. Epub 2014 Oct 7. PMID 25291189
- [Result] Meyer D. Iron chelation as therapy for HIV and Mycobacterium tuberculosis co-infection under conditions of iron overload. Curr Pharm Des. 2006;12(16):1943-7. doi: 10.2174/138161206777442164. PMID 16787239
- [Result] Cinatl J, Scholz M, Weber B, Cinatl J, Rabenau H, Markus BH, Encke A, Doerr HW. Effects of desferrioxamine on human cytomegalovirus replication and expression of HLA antigens and adhesion molecules in human vascular endothelial cells. Transpl Immunol. 1995 Dec;3(4):313-20. doi: 10.1016/0966-3274(95)80017-4. PMID 8665150
- [Result] Mabeza GF, Loyevsky M, Gordeuk VR, Weiss G. Iron chelation therapy for malaria: a review. Pharmacol Ther. 1999 Jan;81(1):53-75. doi: 10.1016/s0163-7258(98)00037-0. PMID 10051178
- [Result] Weinberg GA. Iron chelators as therapeutic agents against Pneumocystis carinii. Antimicrob Agents Chemother. 1994 May;38(5):997-1003. doi: 10.1128/AAC.38.5.997. PMID 8067783
- [Result] Paradkar PN, De Domenico I, Durchfort N, Zohn I, Kaplan J, Ward DM. Iron depletion limits intracellular bacterial growth in macrophages. Blood. 2008 Aug 1;112(3):866-74. doi: 10.1182/blood-2007-12-126854. Epub 2008 Mar 27. PMID 18369153
- [Result] Giannakopoulou E, Pardali V, Zoidis G. Metal-chelating agents against viruses and parasites. Future Med Chem. 2018 Jun 1;10(11):1283-1285. doi: 10.4155/fmc-2018-0100. Epub 2018 May 3. No abstract available. PMID 29719970
- [Result] Gordeuk V, Thuma P, Brittenham G, McLaren C, Parry D, Backenstose A, Biemba G, Msiska R, Holmes L, McKinley E, et al. Effect of iron chelation therapy on recovery from deep coma in children with cerebral malaria. N Engl J Med. 1992 Nov 19;327(21):1473-7. doi: 10.1056/NEJM199211193272101. PMID 1406879
- [Result] Duchemin JB, Paradkar PN. Iron availability affects West Nile virus infection in its mosquito vector. Virol J. 2017 Jun 5;14(1):103. doi: 10.1186/s12985-017-0770-0. PMID 28583206